CLINICAL TRIAL: NCT05225844
Title: Camrelizumab Plus Apatinib Mesylate for Advanced Gastrointestinal Cancer With Previous Standard Treatment Failure ：an Exploratory, Single-arm, Open-label, Phase II Trial
Brief Title: An Exploratory Trail of Camrelizumab Plus Apatinib Mesylate for Advanced Gastrointestinal
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Han, Chief physician, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1-23
Record Dates: First submitted 2022-01-24; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Cancer; Immunotherapy; Targeted Therapy
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab Plus Apatinib mesylate (Experimental): for advanced gastric cancer with previous standard treatment failure
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate
- Camrelizumab and Apatinib mesylate (Experimental): for advanced colorectal cancer with previous standard treatment failure
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab ，200mg/㎡，d1，ivgtt，every 21 days as a cycle
Drug: Apatinib Mesylate — Apatinib Mesylate，250mg/㎡，po，d1-5 on/d2 off，every 21 days as a cycle

SUMMARY:
At present, surgery, radiotherapy and chemotherapy are the main treatment methods for patients with advanced gastrointestinal cancer. Although targeted therapy has significantly improved the prognosis of patients, the mortality of patients has not been significantly reduced, so new treatment methods are urgently needed. In recent years, immunotherapy has become a new hotspot in tumor therapy. Compared with traditional treatment, immune checkpoint inhibitors (ICIS) have shown long-term good efficacy and tolerance in clinical trials. However, single drug ICIS has reached a bottleneck for advanced gastrointestinal cancer, with low response rate and poor PFS and OS. With the results of REGONIVO showing good efficacy, the treatment mode of immune combined with small molecule anti angiogenesis drugs has sprung up. The purpose of this study was to analyze the efficacy and safety of in Camrelizumab combination with Apatinib mesylate in advanced gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed as gastric or colorectal adenocarcinoma by histopathology and/or cytology.

  2. Patients could not receive surgical resection. 3. Previous standard treatment failure . 4. According to the RECIST v1.1 guide, at least 1 lesions (never received radiotherapy),accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) (intravenous contrast agent as the first choice),the longest diameter was more than 10mm (except for the lymph nodes, the short axis of the lymph nodes must be more than 15mm), repeated measurement.

  5.Eastern Cooperative Oncology Group Performance Status(ECOG PS):0-1 score 6.The main organs function is normal, which meets the following requirements. (1) Blood routine examination,(no blood transfusion within 14 days).
  1. Hemoglobin(HB)≥90g/L;
  2. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
  3. Blood platelet (PLT)≥80×10^9/L; (2) Biochemical examination should comply with the following criteria:

  <!-- -->

  1. Bilirubin(BIL) <1.5 times of the upper limit of normal value (ULN)
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase(AST)<2.5*ULN (liver metastasis ALT and AST<5*ULN).
  3. Serum Cr≤1*ULN, creatinine clearance rate≥50ml/min(Cockcroft-Gault formula) 7. The expected survival time more than 3 months; 8. The physicians plan to use Camrelizumab Plus Apatinib Mesylate. 9. Patients voluntarily joined the study and signed informed consent form(ICF). 10. Childbearing age women must undergo a negative pregnancy test(serum or urine) within 7 days ,and voluntarily adopt appropriate methods for contraception from the period of under observation and within 8 weeks of the last time they are given the drug;As for men, it is necessary to receive surgical sterilization, or agree to adopt appropriate methods for contraception from the period of under observation and within 8 weeks of the last time they are given the drug.

Exclusion Criteria:

1. There is a case of heart disease in any of the following situations. (1)Recent publications have the following heart disease (within 6 months)

   1. Acute coronary artery syndrome
   2. Acute heart failure (grade III or IV of NYHA classification)
   3. Significant ventricular arrhythmia(sustained ventricular tachycardia, ventricular fibrillation and sudden death after resuscitation).

      (2)The New York Heart Association(NYHA) grade of grade III or IV (3)The patients with severe conduction block, and permanent pacemaker is invalid (two degree and three degree atrioventricular block, sinus arrest) (4)Unexplained syncope occurred within 3 months.

      (5)The researchers identified as uncontrol of severe hypertension, or symptomatic hypertension.
2. There are many factors that affect the absorption of oral drugs (such as unable to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction).
3. ECOG score≥2
4. Abnormal coagulation function (INR>1.5*ULN, Activated Partial Thromboplastin Time (APTT)>1.5*ULN), with bleeding tendency.
5. There is any history of allergy or hypersensitivity in this research's drug or adjuvant.
6. HIV infection and/or active hepatitis B virus infection.
7. Any condition that may damage the safety of patients or the integrity of research data, including serious medical risk factors, physical condition and laboratory abnormality.
8. The high risk population carrying UGT1A1*28 (7/7) *6 (A/A) genotype or simultaneous carrying of the UGT1A1*28 (6/7) *6 (A/G) genotype (the heterozygous genotype) suggests the exclusion of the Irinotecan
9. Pregnant or lactating women;
10. Other conditions which the doctor think not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  The proportion of patients whose tumor is reduced to a certain amount and maintain a certain period of time.
progression-free survival（PFS） | 24 months
  the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier)

SECONDARY OUTCOMES:
Overall Survival（OS） | 24 months
  overall survival time after the beginning of the treatment
Adverse Events | 24 months
  Adverse events will be evaluated according to NCI CTCAE 4.0
Disease control rate(DCR) | 24 months
  The rate of cases of remission and stable disease accounts for the total evaluable cases after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China